CLINICAL TRIAL: NCT03369717
Title: Use of Perioperative Antibiotics in Endoscopic Sinus Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated early
Sponsor: Montefiore Medical Center (Other)
Collaborators: Mount Sinai Hospital, New York (Other); NYU Langone Health (Other); Weill Medical College of Cornell University (Other); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-8460
Record Dates: First submitted 2017-12-06; First posted 2017-12-12 (Actual); Results first posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Chronic Sinus Infection
Keywords: endoscopic sinus surgery; antibiotics
MeSH Terms: interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Antibiotics (Experimental): To receive postoperative antibiotics
  Interventions: Drug: Amoxi Clavulanate
- No antibiotics (No Intervention): Will not receive any postoperative antibiotics

INTERVENTIONS:
Drug: Amoxi Clavulanate — Postoperative antibiotics
  Arms: Antibiotics

SUMMARY:
The objective of this study is to determine whether the use of postoperative antibiotics following endoscopic sinus surgery (ESS) decreases postoperative infection rates. This is a multi-institutional prospective study involving Albert Einstein College of Medicine/Montefiore Medical Center, Columbia University Medical Center, Weill Cornell Medical College, Mount Sinai Health System, and New York University Langone Medical Center. The study design will be a multi-institutional prospective randomized controlled trial with parallel random groups assigned to receive postoperative antibiotics or no postoperative antibiotics. The investigators hypothesize that patients who receive postoperative antibiotics will have lower postoperative infection rates and improved postoperative sinonasal symptoms and nasal endoscopy scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Chronic Rhinosinusitis (CRS) with or without nasal polyposis or allergic fungal rhinosinusitis who present to the otolaryngology clinic who have been deemed suitable for bilateral ESS, and are over the age of 18 will be included.

Exclusion Criteria:

* Patients with sinonasal tumors, allergies or adverse reactions to all of the antibiotics that will be used in this study (amoxicillin-clavulanate, doxycycline, clarithromycin), immunodeficiency, cystic fibrosis, pregnancy, or diabetes with nasal polyposis (inability to receive systemic steroids) will be excluded, as will patients who lack capacity to provide informed consent. Patients undergoing active treatment for malignancy will be excluded. Patients undergoing unilateral ESS or with nonabsorbable packing placed at the time of surgery will be excluded. Patients who have been on antibiotics within 2 weeks of the surgery date will be excluded. Patients with acute on chronic sinusitis or the presence of purulence at time of surgery will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2020-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadeem Akbar, MD, Principal Investigator — Assistant Professor
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Antibiotics | No Antibiotics
Started | 12 | 12
Completed | 2 | 4
Not Completed | 10 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Antibiotics | No Antibiotics | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 18
  >=65 years | 2 | 4 | 6
Age, Continuous [Mean (Full Range); unit: Years] | 52 [25 to 71] | 46 [22 to 74] | 49 [22 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 7 | 4 | 11
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 7 | 4 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Active Infection at time of surgery [Count of Participants; unit: Participants] — The number of participants with an active infection at the time of surgery is summarized by study arm.
  Participants | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Infection
Description: The number/percentage of participants with postoperative infection rate, as assessed by rigid nasal endoscopy in the office and culture of suspected infectious material noted within the paranasal sinuses will be reported. A postoperative infection as defined by having an infection at ANY of the postoperative visits AND detected initially by evidence of purulence on nasal endoscopy will be considered an infection if the culture swab from the site of purulence during that office visit confirms that there is an actual bacterial source of the infection.
Time Frame: During all three scheduled postoperative visits: 7-10 days postoperatively; 2-4 weeks postoperatively; 6-8 weeks postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotics | No Antibiotics
Number analyzed (Participants) | 12 | 12
Participants | 1 | 0

2. Secondary Outcome: Postoperative Sino-nasal Outcome Test (SNOT-22) Scores
Description: Postoperative SNOT-22 scores will be summarized for each visit based on patient-reported symptoms. The SNOT-22 is a 22-item questionnaire used to assess the impact of chronic rhinosinusitis (CRS) on a patient's health-related quality of life. Participants are presented with a list of symptoms and social/emotional consequences of rhinosinusitis and asked to rate each problem over the prior 2-week period on a 6-point Likert scale ranging from 0 ("No Problem") to 5 ("Problem as bad as it can be)" yielding an overall possible scoring range of 0-110. Higher scores are indicative of a greater burden CRS-related symptoms. Scores are summarized by study arm using basic descriptive statistics.
Time Frame: as for outcome 1
Population: The numbers reflect loss of follow up of patients during successive visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Antibiotics | No Antibiotics
Number analyzed (Participants) | 12 | 12
score on a scale
  7 to 10 days post op | 25 (2) | 22 (1)
  2 to 4 weeks post op: number analyzed (Participants) | 8 | 10
  2 to 4 weeks post op | 23 (1.5) | 21 (0.5)
  6 to 8 weeks post op: number analyzed (Participants) | 2 | 4
  6 to 8 weeks post op | 22 (0.5) | 21 (0.5)

3. Secondary Outcome: Perioperative Sinus Endoscopy (POSE) Scores
Description: Sinonasal crusting and inflammation was determined using the perioperative sinus endoscopy (POSE) scoring system based on patient-reported symptoms obtained during all three study visits. POSE assigns points to various areas within the nasal passages, based on the presence of certain conditions like crusting, edema, polyps, secretions, etc. For purposes of this study each parameter was scored from 0-2 yielding an overall possible score of 0-10, with higher scores being indicative of more extensive disease severity or surgical extent in the sinuses. Scores are summarized by study arm using basic descriptive statistics.
Time Frame: as for outcome 1
Population: The numbers reflect loss of follow up of patients during successive visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Antibiotics | No Antibiotics
Number analyzed (Participants) | 12 | 12
score on a scale
  7 to 10 days post op | 5.4 (1.4) | 5.2 (1.1)
  2 to 4 weeks post op: number analyzed (Participants) | 8 | 10
  2 to 4 weeks post op | 4.3 (0.6) | 4.1 (0.8)
  6 to 8 weeks post op: number analyzed (Participants) | 2 | 4
  6 to 8 weeks post op | 3.8 (0.2) | 3.5 (0.4)

ADVERSE EVENTS:
Time Frame: Up to 8 weeks following endoscopic sinus surgery
Arm/Group | Antibiotics | No Antibiotics
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
We had a very low enrollment and therefore were unable to reach any statistical significance with any of our endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-27): https://cdn.clinicaltrials.gov/large-docs/17/NCT03369717/Prot_SAP_000.pdf